CLINICAL TRIAL: NCT04053088
Title: Surgical Aortic Valve Replacement: IMPACT of Pre-existing Comorbidities on Patient Outcomes and Prosthetic Valve Performance in a Real-world Setting.
Brief Title: SAVR: IMPACT of Pre-existing Comorbidities on Patient Outcomes and Prosthetic Valve Performance in a Real-world Setting.
Acronym: IMPACT
Status: Active, not recruiting | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: IPPM2019IMPACT
Record Dates: First submitted 2019-08-06; First posted 2019-08-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases
Keywords: Surgical Aortic Valve Replacement (SAVR); INSPIRIS RESILIA; Durability; Hemodynamics
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SAVR patients: patients undergoing surgical aortic valve replacement (SAVR) by usage of the INSPIRIS RESILIA Aortic valve™
  Interventions: Device: INSPIRIS RESILIA Aortic Valve™

INTERVENTIONS:
Device: INSPIRIS RESILIA Aortic Valve™ — Collection of patient data from patients undergoing Surgical Aortic Valve Replacement (SAVR) by usage of the INSPIRIS RESILIA aortic valve™

SUMMARY:
The IMPACT Registry represents a non-interventional, prospective, open-label, multicenter, international registry with a follow-up of 5 years that includes data of patients undergoing aortic valve replacement with the Edwards INSPIRIS RESILIA Aortic Valve™. The IMPACT Registry will be performed in up to 25 participating sites across Germany, Austria and Switzerland. A minimum number of 500 patients (20 patients per center) will be enrolled. Patients will undergo follow-up visits at baseline, surgery, pre-discharge, year 1, year 3 and year 5.

DETAILED DESCRIPTION:
The INSPIRIS RESILIA Aortic Valve™ is a stented tri-leaflet valve comprised of bovine pericardial tissue. The tissue is created by treating bovine pericardial tissue with Edwards Integrity Preservation. It incorporates a stable capping anticalcification process, which blocks residual aldehyde groups known to bind with calcium. Tissue preservation with glycerol allows the valve to be stored without a traditional liquid-based solution, such as glutaraldehyde. Therefore, valve is stored under dry packaging conditions and consequently does not require rinsing prior to implantation.

The novel tissue preservation technology significantly improves hemodynamic and anticalcification properties compared with the standard Perimount valve in an ovine model (Flameng et al., 2015). The RESILIA tissue has been studied in the COMMENCE trial: Two year data show that the NYHA class improved in 65.7% of patients, effective orifice area after implantation was 1.6 ± 0.5 cm2; mean gradient was 10.1 ± 4.3 mmHg; and paravalvular leak was none/trivial in 94.5% of patients (mild to moderate in 0.5%) (Puskas et al., 2017).

On the sizes 19 - 25 mm the INSPIRIS RESILIA Aortic Valve™ has been outfitted with the VFit technology, which incorporates two novel features designed for potential future valve-in-valve procedures: fluoroscopically visible size markers and an expandable cobalt chromium alloy band. No clinical data are available that evaluate the use of the INSPIRIS RESILIA Aortic Valve™ in patients to date.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years old
2. Patient has an aortic valve vitium and requires an aortic valve replacement with the Edwards INSPIRIS RESILIA Aortic Valve™
3. Patient is scheduled to attend yearly follow-up visits at the registry center up to 5 years
4. Patient provides written informed consent prior to the procedure and in case of emergency after the procedure.

Exclusion Criteria:

1. Disability and / or other circumstances under which the patient is not capable to understand the nature, significance and scope of the clinical trial
2. Active endocarditis/myocarditis or endocarditis/myocarditis within 3 months prior to the scheduled aortic valve replacement surgery
3. Patient has a life expectancy ≤ 12 months for any reason
4. Valve implantation is not possible in accordance with the device IFU
5. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Minimum of 500 patients (20 patients per center) undergoing Surgical Aortic Valve Replacement (SAVR) using the INSPIRIS RESILIA aortic valve™ (all comers).
  The required sample size was calculated using the online calculator at http://www.surveysystem.com/sscalc.htm. It was estimated, from the COMMENCE Trial dataset (Puskas et al., 2017) that all-cause mortality is around 1.2% at year 1 and 2.0% at year 2.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | after 1 year
  All-cause mortality after 1 year will be investigated
All-cause mortality | after 3 years
  All-cause mortality after 3 years will be investigated
All-cause mortality | after 5 years
  All-cause mortality after 5 years will be investigated

SECONDARY OUTCOMES:
Mortality | after 1 year
  All cause, cardiac and valve-related mortality in the overall study population and in different patient subgroups at all timepoints: Chronic kidney disease, diabetes, hypertension, metabolic syndrome, inflammation
Mortality | after 3 years
  All cause, cardiac and valve-related mortality in the overall study population and in different patient subgroups at all timepoints: Chronic kidney disease, diabetes, hypertension, metabolic syndrome, inflammation
Mortality | after 5 years
  All cause, cardiac and valve-related mortality in the overall study population and in different patient subgroups at all timepoints: Chronic kidney disease, diabetes, hypertension, metabolic syndrome, inflammation

OTHER OUTCOMES:
Change in Maximum pressure gradient (Pmax) over time | after 1 year
  Change in Pmax in mmHg as an indicator of patient prosthesis mismatch
Change in Maximum pressure gradient (Pmax) over time | after 3 years
  Change in Pmax in mmHg as an indicator of patient prosthesis mismatch
Change in Maximum pressure gradient (Pmax) over time | after 5 years
  Change in Pmax in mmHg as an indicator of patient prosthesis mismatch
Change in mean pressure gradient (Pmean) over time | after 1 year
  Change in Pmean in mmHg as an indicator of patient prosthesis mismatch
Change in mean pressure gradient (Pmean) over time | after 3 years
  Change in Pmean in mmHg as an indicator of patient prosthesis mismatch
Change in mean pressure gradient (Pmean) over time | after 5 years
  Change in Pmean in mmHg as an indicator of patient prosthesis mismatch
Change in velocity time integral (VTI) over time | after 1 year
  Change in VTI as an indicator of patient prosthesis mismatch
Change in velocity time integral (VTI) over time | after 3 years
  Change in VTI as an indicator of patient prosthesis mismatch
Change in velocity time integral (VTI) over time | after 5 years
  Change in VTI as an indicator of patient prosthesis mismatch
Change in prostesis opening area (EOA) over time | after 1 year
  Change in EOA in mm2 as an indicator of patient prosthesis mismatch
Change in prostesis opening area (EOA) over time | after 3 years
  Change in EOA in mm2 as an indicator of patient prosthesis mismatch
Change in prostesis opening area (EOA) over time | after 5 years
  Change in EOA in mm2 as an indicator of patient prosthesis mismatch
Change in left ventricular ejection fraction (LVEF) over time | after 1 year
  Change in LVEF in % as an indicator of patient prosthesis mismatch
Change in left ventricular ejection fraction (LVEF) over time | after 3 years
  Change in LVEF in % as an indicator of patient prosthesis mismatch
Change in left ventricular ejection fraction (LVEF) over time | after 5 years
  Change in LVEF in % as an indicator of patient prosthesis mismatch
Occurence of paravalvular leaks | after 1 year
  Occurence of paravalvular leaks as an indicator of patient prostheis mismatch
Occurence of paravalvular leaks | after 3 years
  Occurence of paravalvular leaks as an indicator of patient prostheis mismatch
Occurence of paravalvular leaks | after 5 years
  Occurence of paravalvular leaks as an indicator of patient prostheis mismatch
Occurence of structural valve detioration (SVD) over time | after 1 year
  SVD to be determined by imaging methods (e.g. Echocardiography) following Salaun et al. 2018
Occurence of structural valve detioration (SVD) over time | after 3 years
  SVD to be determined by imaging methods (e.g. Echocardiography) following Salaun et al. 2018
Occurence of structural valve detioration (SVD) over time | after 5 years
  SVD to be determined by imaging methods (e.g. Echocardiography) following Salaun et al. 2018
Occurence of repeat procedures (valve-in-valve reoperation) | after 1 year
  Any repeat procedures will be documented and assessed
Occurence of repeat procedures (valve-in-valve reoperation) | after 3 years
  Any repeat procedures will be documented and assessed
Occurence of repeat procedures (valve-in-valve reoperation) | after 5 years
  Any repeat procedures will be documented and assessed
New York Heart Association (NYHA) functional class compared to baseline | after 1 year
  NYHA class will be determined at follow-up visits
New York Heart Association (NYHA) functional class compared to baseline | after 3 years
  NYHA class will be determined at follow-up visits
New York Heart Association (NYHA) functional class compared to baseline | after 5 years
  NYHA class will be determined at follow-up visits
Freedom from valve-related rehospitalization | after 1 year
  any valve related hospitalizations will be documented and assessed
Freedom from valve-related rehospitalization | after 3 years
  any valve related hospitalizations will be documented and assessed
Freedom from valve-related rehospitalization | after 5 years
  any valve related hospitalizations will be documented and assessed
Need for new pacemaker implant | after 1 year
  Any occurence of new pacemaker implant (e. g. when the participant did not have a pacemaker at baseline) will be documented and assessed
Need for new pacemaker implant | after 3 years
  Any occurence of new pacemaker implant (e. g. when the participant did not have a pacemaker at the preceding follow-up visit) will be documented and assessed
Need for new pacemaker implant | after 5 years
  Any occurence of new pacemaker implant (e. g. when the participant did not have a pacemaker at the preceding follow-up visit) will be documented and assessed

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Bakhtiary, Dr. med., Principal Investigator — Helios Klinik Siegburg; Andreas Zierer, Prof. Dr., Principal Investigator — Kepler University Hosiptal Linz and Hospital Wels-Grieskirchen
Locations (22):
- Austria (4):
  - Medizinische Universität Innsbruck, Uniklinik für Herzchirurgie, Innsbruck
  - Kepler Universitätsklinikum Linz, Linz
  - • Universitätsklinikum Salzburg, Herzchirurgie, Gefäßchirurgie und endovaskuläre Chirurgie, Salzburg
  - • Klinikum Wels-Grieskirchen, Herz-, Gefäß- und Thoraxchirurgie, Wels
- Germany (15):
  - Klinikum Nürnberg, Nuremberg, Bavaria
  - Klinikum Passau/Universität Regensburg, Passau, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - • Universitätsklinikum Frankfurt, Thorax-, Herz- und thorakale Gefässchirurgie, Frankfurt am Main, Hesse
  - Universitätsklinik für Herzchirurgie, Oldenburg, Lower Saxony
  - Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia
  - Schüchtermann Klinik, Bad Rothenfelde, North Rhine-Westphalia
  - Herzzentrum Bergmannsheil, Bochum, North Rhine-Westphalia
  - Klinik für Herzchirurgie UKD, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - • Universitätsklinikum Leipzig, Thorax- und Kardiovaskuläre Chirurgie, Leipzig, Saxony
  - BundeswehrKrankenhaus Klinik XVII und XVIII, Koblenz
  - Helios Klinikum Siegburg, Siegburg
  - Universitätsklinikum Ulm, Ulm
  - Helios Klinikum Wuppertal, Wuppertal
- Catharina Ziekenhuis, Catharina Hart- en Vaatcentrum, Eindhoven, Netherlands
- Switzerland (2):
  - HerzKlinik Hirslanden, Herz- und thorakale Gefässchirurgie, Zurich
  - HerzZentrum Hirslanden, Herz- und Gefässchirurgie, Zurich

REFERENCES:
- [Background] Salaun E, Clavel MA, Rodes-Cabau J, Pibarot P. Bioprosthetic aortic valve durability in the era of transcatheter aortic valve implantation. Heart. 2018 Aug;104(16):1323-1332. doi: 10.1136/heartjnl-2017-311582. Epub 2018 May 7. PMID 29735584
- [Derived] Bakhtiary F, Ahmad AE, Autschbach R, Benedikt P, Bonaros N, Borger M, Dewald O, Feyrer R, Geissler HJ, Grunenfelder J, Lam KY, Leyh R, Liebold A, Czesla M, Mehdiani A, Pollari F, Salamate S, Strauch J, Votsch A, Weber A, Wendt D, Botta B, Bramlage P, Zierer A. Impact of pre-existing comorbidities on outcomes of patients undergoing surgical aortic valve replacement - rationale and design of the international IMPACT registry. J Cardiothorac Surg. 2021 Mar 25;16(1):51. doi: 10.1186/s13019-021-01434-w. PMID 33766089